CLINICAL TRIAL: NCT05261906
Title: The Libre Enabled Reduction of A1c Through Effective Eating and Exercise Study: LIBERATE
Brief Title: The FreeStyle Libre Enabled Reduction of A1c Through Effective Eating and Exercise Study
Acronym: LIBERATE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: Abbott Diabetes Care (Industry)
Responsible Party: Principal Investigator, Sonja Reichert, Associate Professor, Department of Family Medicine; Dr. Brian W. Gilbert Chair in Primary Health Care Research, Western University, Canada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 119334
Record Dates: First submitted 2022-01-27; First posted 2022-03-02 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: lifestyle medicine; flash glucose monitor; exercise prescription; nutrition; biofeedback; self-monitoring; wearable activity monitor; virtual care; group education; coaching; behaviour change
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: All participants will be in the treatment group. This is a multisite intervention; the intervention will be first delivered at the Primary Care for Diabetes Support Program in London, Ontario with 92 participants. Following intervention completion in London, ON, the Boris Clinic in Diabetes Care and Research Program (DCRP) in Hamilton, ON will deliver the intervention as a fidelity check, with another 92 participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LIBERATE Intervention (Experimental)
  Interventions: Behavioral: LIBERATE

INTERVENTIONS:
Behavioral: LIBERATE — Five bi-weekly, followed by three monthly, one-hour videoconferencing group education classes via Microsoft Teams video platform will be offered. Participants will be given the choice to communicate with the LIBERATE clinical team (exercise specialist, MD, and/or RN) weekly between the group classes using their preferred method of communication i.e., email.
  Classes will offer FreeStyle® Libre-assisted behavioural coaching (i.e., nutrition and exercise). FreeStyle® Libres will be used during the first three months of the program and optionally in the last three months of the intervention. The FitBit Inspire 2™ monitors will be worn for six months. Participants are provided the option to receive individualized aerobic and resistance training prescriptions.

SUMMARY:
This two-year multisite, real-world, before-after prospective six-month pilot study utilizing a single-group cohort design (n=184) which will first occur in London, Ontario (n=92) through the St. Joseph's Primary Care for Diabetes Support (PCDSP) program. To test fidelity, the intervention will be delivered again in Hamilton, Ontario through the Hamilton Health Sciences' Boris Clinic in Diabetes Care and Research Program (n=92).

Participants will begin by attending the first class at the PCDSP clinic to complete baseline fitness testing as well as receive/set up their wearable technology (FitBit Inspire 2™ and FreeStyle® Libre sensors). Two weeks of baseline data collection will following (glucose values and step counts). Five bi-weekly, followed by three monthly, one-hour videoconferencing group education classes via Microsoft Teams video platform will be offered. Participants will be given the choice to communicate with the LIBERATE clinical team (exercise specialist, physician, and/or registered) weekly between the group classes using their preferred method of communication i.e., email.

Classes will offer FreeStyle® Libre-assisted behavioural coaching (i.e., nutrition and exercise). FreeStyle® Libres will be used during the first three months of the program and optionally in the last three months of the intervention. The FitBit Inspire 2™ monitors will be worn for six months. Participants are provided the option to receive individualized aerobic and resistance training prescriptions. The primary outcome is change in glycated hemoglobin. A main goal of this study is to create a "toolkit" for other Canadian Diabetes Management centres (DMCs) to use in the future.

DETAILED DESCRIPTION:
PROTOCOL TIMELINE

A. Pre-study Eligibility Criteria Confirmation and Study Review and Scheduling of Participant

The research coordinator will phone potential participants to answer any questions about the study and confirm eligibility criteria. One the same call, the research coordinator will be setting up a phone call time (within the week) to review the LOI with the potential participant. After the phone call, the research coordinator will send the LOI for review via email. The time from this call to program start may vary between participants. This is due to the need to fill the group capacity of 6-8 participants/class before initiating a participant.

If a patient self-refers from the community, we will access OLIS for recent blood work. If an A1c has not been completed in the last 3 months, we will need to consent them over the phone using the e-consent via REDCap first and then they will be given an OHIP lab requisition to complete the test within one week. This is done so that potential participants are not having to go through the entire onboarding testing before knowing if they are eligible to participate in the study.

On the phone call (within the week of the pre-screening call), we will review the Letter of Information and Consent with the participant. We will answer any questions they may have.

B. Time 1: ORIENTATION SESSION

The first group session will hopefully be in-person. If however we are unable to do so, we will use the WebEx platform to orient and teach participants about the technology they will be using during the study. This session will be run by a CDNE and the research coordinator.

We will review study expectations briefly at the session, answer any remaining questions about the LOI. Then, informed consent will be obtained virtually using individualized REDCap links to sign the board approved e-consent method.

Topics to be covered during this session will include; how to set-up and use the wearable fitness tracker (FitBit Inspire 2™) and FreeStyle® Libre, and their associated smartphone apps. To ensure safety to participate in exercise, the modified Physical Activity Readiness Questionnaire (PAR-Q) will also be administered by either and RN or MD at this time (Freehan et al., 2018). If they pass the PAR-Q, baseline fitness testing (see "other measures section" for description of the six-minute walk test (6MWT) and handgrip testing protocol) will also occur during this session. Participants will also complete their baseline stride length assessment, weight, and height, blood pressure and waist circumference assessments. Baseline questionnaires will be completed via online surveys.

Once consent is obtained, and medical suitability is confirmed baseline physiological data (glycated hemoglobin (HbA1c), medications, past medical history) will be extracted from the PCDSP electronic medical record (EMR) WebDR. If the patient is referred to us by a family physician we will ask them to include these details in the referral.

C. Intervention Week 1-12 (IW2-12): Biweekly Virtual Sessions

* Within Intervention week 1, participants will be randomly prompted to complete a 24h-hour dietary recall through the ASA-24 2018, completed 3 times within the week. All participants will complete this measurement; each participant will be assigned to a random day within the week to avoid planning healthy meals (and creating biased results).
* Baseline Step Count and FreeStyle Libre Data Collection (2 weeks) after attending the on-boarding session

Then after the two week baseline, participants will attend biweekly virtual coaching sessions (total of six (6) classes including the on-boarding session). Please see below for an outline of the proposed content delivered during the classes (coaching program: behavioural, nutrition and exercise). Prior to each virtual group i.e. the night before, participants will be required to email: 1) wearable fitness tracker data (screen shot of their exercise/step summary), 2) resistance training log if engaging with resistance exercise as a method of glucose regulation and 3) uploaded sensor data to LibreView. This information will then be reviewed by a clinic exercise specialist/registered nurse/ physician prior to the group to determine individualized exercise progression, and suggested modifications to diet. Wearable fitness study-related data will NOT be collected via these means (email), but rather via data export from the fitbit.com desktop platform completed by the research co-ordinator. Participants will provide us an email address to use on their behalf, and we will provide a password for participants to use to log on to their smartphone app (or desktop platform, if they wish) during the course of the study. After the study, participants will be granted permission to change their password to a desired password, and study investigators will lose access to this account.

At the end of the 12 weeks, participants will be asked to go have their blood tested within (given a blood requisition for A1c testing). They will also be asked to come into the clinic to have their weight, height, and waist circumference measured. Participants will also re-complete the 6MWT and handgrip strength test. At the same time, participants will be given their final three FreeStyle Libre 2 sensors.

Within Intervention week 12, participants will be randomly prompted to complete a 24h-hour dietary recall through the ASA-24 2018, three times within the week. All participants will complete these measurements; each participant will be assigned to a random day within the week. When prompted via email, participant will be asked to complete a recall of the past day from midnight to midnight of all that they ate and drank.

D. Intervention Week 12-24 (IW12-24): Monthly Virtual Sessions Coaching during the remaining 3 virtual group education classes (on Microsoft Teams) of the last 3 months of the intervention will be similar in design to IW2-12, but will focus on creating lasting behaviour change. Participants will be given the choice whether to wear any or all of their three (3) Libre 2 sensors and/for continue to wear the loaned FitBit Inspire 2™. Sensor usage will be tracked (i.e., Participant 3 used 2/3 sensors).

E. Follow-up Period (Week 24) Participants will be contacted to set up an appointment to review the follow-up questionnaires in clinic with the research coordinator. The questionnaires to be completed are: the Stanford Diabetes Self-Efficacy Scale, EQ-5D-5L, and an exit survey. Participants will also return the FitBit Inspire 2™ back to the clinic. Participants will also attend their fitness testing (6MWT and handgrip strength test) at the clinics. Participants will receive a A1c requisition again to have A1c tested again within the week.

Within Intervention week 24, participants will be randomly prompted to complete a 24h-hour dietary recall through the ASA-24 2018, completed 3 times within the week. All participants will complete this measurement; each participant will be assigned to a random day within the week. When prompted via email, participant will be asked to complete a recall of the past day from midnight to midnight of all that they ate and drank.

Intervention Description:

A. Intervention Week 2-12 (IW2-12): Biweekly Virtual Sessions

Participants will attend biweekly virtual coaching sessions (total of five (5) classes). Prior to each virtual group i.e. the night before, participants will be required to email: wearable fitness tracker information (resistance exercise log if applicable) and uploaded sensor data to LibreView. This information will be reviewed by a clinic registered nurse or physician prior to the group to determine individualized exercise progression, and suggested modifications to diet.

B. Intervention Week 12-24 (IW12-24): Monthly Virtual Sessions

Coaching during the remaining 3 classes of the last 3 months of the intervention will be similar in design to IW2-12, but will focus on creating lasting behaviour change. Participants will be given the choice whether or not to wear any or all of their three (3) Libre sensors.

C. Coaching Program Description

At the beginning of each class, participants will be given their new exercise AND nutrition goal or prescription. For the remainder of the 1-hour class, the focus will be to coach participants to infer and draw connections between their food/activity choices and glycemic responses. This will be done using motivational interviewing guided by Self Determination Theory and Kolb's cycle of experiential learning and Libre glycemic examples from volunteering participants. Participants will be encouraged to have their Libre results from the previous two weeks in front of them to use during these exercises. Focusing on habit formation will also be a key coaching goal.

Participants will for the most part lead the direction of the group discussion, with questions raised at the start of each session by the group facilitator(s): barriers or motivators in the last two weeks, goals achieved, etc. The clinical group facilitators coaching the group will provide suggestions or solutions to issues i.e. technology issues, how to safely exercise in a pandemic environment, how to reduce glycemic variability by choosing lower glycemic foods, etc. Didactic teaching will be kept to a minimum to optimize adult learning behaviour and theory.

D. FreeStyle Libre Assisted Nutrition Coaching Description

Focus of the material presented during these classes will be to guide participants towards the consumption of lower carbohydrate and lower glycemic foods, while maintaining adequate nutritional needs for activity and health. General principles will be provided at the start of the program, with participants then learning, based on their FreeStyle Libre glycemic readings which foods affect their blood sugars in both positive and negative ways. The goal will be to empower participants to not only find day-to-day foods that work for their diabetes, but also to be able to critically evaluate food choices when the foods consumed either raise or lower blood sugars to undesired levels.

E. Exercise Prescriptions

Step, aerobic and resistance training prescriptions will be updated biweekly for baseline-month 3 (within one day of group classes) and will continue on the same schedule (biweekly) after month 3 to month 6.

Participants will be encouraged to interrupt their prolonged sitting with frequently (every 20 to 45 minutes, under an hour) with 2-3 minutes light-intensity physical activity and to decrease overall daily sedentary time. To give participants daily feedback and reminders to get up and move every hour, participants are advised to achieve their hourly movement goals (defined as an hour with 250 steps or more, defined and measured by the FitBit Inspire 2™) or 2 to 3 minutes of light physical activity.

ELIGIBILITY:
Inclusion Criteria:

- • Diagnosis of Type 2 diabetes, age >18 years old

* Baseline HbA1c ≥ 8.0% (if no recent A1c (last 3 months) you can ask, or we will ask them to complete a new test).
* Naïve to Flash glucose monitors BUT interested in using this technology
* Ownership of either a smartphone (iPhone v7 (iOS of 13.2+) or Samsung Galaxy Note 8, S7 Edge, S8, S8+, S9, S10; Google Pixel, Pixel 2, Pixel 2 XL, Pixel 3, Pixel 3 XL, Pixel 4, Pixel 4 X; LG Nexus 5X (with Android OS of 8 or higher). Other smartphones may be compatible but must be confirmed. https://freestyleserver.com/Payloads/IFU/2022/q2/ART39109-002_rev-J-web.pdf
* Have an email address
* Access to Internet connection
* Physician cleared to participate in exercise

Exclusion Criteria:

* • Lack of access/knowledge of technology that would prevent virtual participation (Self-reported)

  * • Language barrier, severe mental illness, cognitive impairment or significant/unstable psychiatric disease limiting group participation
  * Pregnancy
  * Active or untreated conditions that would preclude the safe participation of exercise i.e., foot ulcer, CVD, uncontrolled HTN, retinopathy, etc.
  * Recent (<3 months) medically unstable condition i.e., recent MI, stroke, hospitalization, etc.
  * Inability to participate in the full program (e.g., upcoming surgery, relocating, etc.…)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c from Baseline | 6 months
  HbA1c measured at baseline, 3 months, and 6 months

SECONDARY OUTCOMES:
Change in total daily basal insulin use from baseline | 6 months
  Daily basal insulin use, measured at baseline, 3 months, and 6 months
Change in rapid insulin use from Baseline | 6 months
  Rapid insulin use, measured at baseline, 3 months, and 6 months

OTHER OUTCOMES:
Change in sulfonylurea use from Baseline | 6 months
  Sulfonylurea use, measured at baseline, 3 months, and 6 months
Change in Average minutes per day of time out of range from Baseline | This will be measured and evaluated continuously bi-weekly for the duration of the 6 month study while subjects are using the FreeStyle Libre sensor
  Measured by the FreeStyle Libre sensor
Change in Estimated A1c from baseline | This will be measured and evaluated continuously bi-weekly for the duration of the 6 month study while subjects are using the FreeStyle Libre sensor
  Measured by the FreeStyle Libre sensor
Change in Number of Scans within a 24-hour period from baseline | This will be measured and evaluated continuously bi-weekly for the duration of the 6 month study while subjects are using the FreeStyle Libre sensor
  Measured by the FreeStyle Libre sensor
Average minutes per day of time in range from baseline | This will be measured and evaluated continuously bi-weekly for the duration of the 6 month study while subjects are using the FreeStyle Libre sensor
  Measured by the FreeStyle Libre sensor
Change in Percent Sensor Capture from baseline | This will be measured and evaluated continuously bi-weekly for the duration of the 6 month study while subjects are using the FreeStyle Libre sensor
  Measured by the FreeStyle Libre sensor
Change in Diabetes Status | This will be evaluated at 6 months.
  Looking for an A1c reduction to below <6.5% (remission)
Anthropometric: Change in Weight from baseline | 6 months
  in kilograms, measured at baseline, 3 months, and 6 months
Anthropometric: Change in Height from baseline | 6 months
  in centimeters, measured at baseline, 3 months, and 6 months
Anthropometric: Change in Waist circumference from baseline | 6 months
  in cm, measured at baseline, 3 months, and 6 months
Fitness Capacity: change in Six Minute Walk Test score from baseline and 3 months | 6 months
  The six-minute walking test (6MWT) has been used in populations with T2D and is a validated (Nolen-Doerr et al., 2018) measure of estimated aerobic exercise capacity. The test is a practical, sub-maximal test that ideally requires a 30m corridor or track to be completed (with markings at least every 3 metres). However, the shorter the travelling distance results in less distance completed in the six-minutes due to time taken to reverse directions (American Thoracic Society, 2002). Participants are able to stop whenever and use walking aids if they wish (Regensteiner, 2004).
Fitness Capacity: Change in Handgrip Strength Test score from baseline and 3 months | 6 months
  Long standing diabetes has been linked to significantly lower grip strength (which is an overall indicator of full body strength and risk of mortality) compared to healthy individuals (Ezema et al., 2012; Sayer et al., 2005). This will be assessed using the Southampton Protocol
Psychological: Change in Health-related Quality of Life score from baseline | 6 months
  EQ-5D-5L
Psychological: Change in Diabetes Self Efficacy score from baseline | 6 months
  Stanford Diabetes Self-efficacy scale (Lorig et al., 2009)
Psychological: Change in Intrinsic Motivation for Exercise scores from baseline | 6 months
  Behavioural Regulation in Exericse Questionnaire BREQ-3 (Markland and Tobin (2004) and Wilson et al. (2006)
Change in Step count from baseline | 6 months
  Bi-weekly mean of daily step count; measured by the FitBit Inspire 2™, measured at baseline, 3 months, and 6 months
Change in Sedentary Time from baseline | 6 months
  Bi-weekly mean of sedentary time in minutes; measured by the FitBit Inspire 2™, measured at baseline, 3 months, and 6 months
change in Light Physical Activity from baseline | 6 months
  Bi-weekly mean of light physical activity in minutes; measured by the FitBit - Inspire 2™; measured at baseline, 3 months, and 6 months
Change in Moderate Physical Activity from baseline | 6 months
  Bi-weekly mean of moderate physical activity in minutes; measured by the FitBit Inspire 2™, measured at baseline, 3 months, and 6 months
Change in Vigorous Physical Activity from baseline | 6 months
  Bi-weekly mean of vigorous physical activity in minutes; measured by the FitBit Inspire 2™, measured at baseline, 3 months, and 6 months
Change in Nutrition (ASA-24) scores from baseline and 3 months | Baseline - 6 months
  ASA-24 Canada Survey.- used to reflect the Canadian food supply, portion sizes, and nutrient composition.
Participant Feedback | Assessed at 6 months
  Assessed using an Exit Survey: completed at the end of the study, to receive feedback about experience/improvements etc.

CONTACTS AND LOCATIONS:
Overall Officials: Sonja M Reichert, MD, Principal Investigator — Western University
Locations (1):
- St. Joseph's Family Medical and Dental Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No